CLINICAL TRIAL: NCT01267266
Title: A Randomized Discontinuation Phase 2 Study of AZD0530 as a Metastasis Inhibitor in Castrate Resistant Prostate Cancer
Brief Title: Saracatinib in Treating Patients With Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Per protocol, study was terminated due to low rate of randomized patients.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02563; NCI-2011-02563 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000691725; 10-436-B (Other: University of Chicago); 8446 (Other: CTEP); N01CM00099 (NIH); N01CM00071 (NIH); U01CA062491 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2010-12-24; First posted 2010-12-28 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2013-01

CONDITIONS: Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — saracatinib; Hydrocortisone

ARMS (2):
- Arm I (saracatinib) (Experimental): Patients receive oral saracatinib once daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: saracatinib
- Arm II (placebo) (Placebo Comparator): Patients receive oral placebo once daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Upon progression, patients may crossover to arm I.
  Interventions: Other: hydrocortisone/placebo

INTERVENTIONS:
Drug: saracatinib — Given orally
  Other Names: AZD0530
  Arms: Arm I (saracatinib)
Other: hydrocortisone/placebo — Given orally
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase II clinical trial is studying how well saracatinib works in treating patients with prostate cancer. Saracatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if AZD0530 (saracatinib) increases time to radiographic progression in men with CRPC compared to placebo.

SECONDARY OBJECTIVES:

I. Describe the adverse events related to AZD0530 in this population. II. Explore the role of FYN and other SRC kinase expression as a predictor of response to AZD0530.

OUTLINE: This is a multicenter study.

LEAD-IN PHASE: Patients receive oral saracatinib once daily during for 8 weeks. Patients who achieve disease regression or a PSA decrease of > 50% continue to receive open-label saracatinib. Patients who do not show radiographic evidence of new metastases on bone scan and CT, disease regression, or a > 50% decrease in PSA continue on to the randomized phase.

RANDOMIZED PHASE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral saracatinib once daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive oral placebo once daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Upon progression, patients may crossover to arm I.

Tissue samples may be collected for correlative studies. After completion of study treatment, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed prostate cancer with progressive disease; progressive disease may be defined as either

  * New clinical or radiographic metastases
  * Rising PSA: PSA must be greater than 1.0 ng/mL with at least 2 consecutive rises after completion of prior therapy; the PSA values documenting these rises should be separated by no less than 10 days; the baseline PSA value may be taken from the end of prior therapy
* Previous treatment with docetaxel for disease progression following hormonal therapy (i.e., castrate-resistant disease) required

  * Treatment in the adjuvant or neoadjuvant setting will NOT be grounds for inclusion unless docetaxel has been used again in the setting of progressive CRPC
* ECOG performance status 0-1
* ANC ≥ 1,500/mm³
* Hemoglobin > 9.0 g/dL
* Platelet count > 100,000/mm³
* Total bilirubin < 2.0 x institutional ULN
* AST/ALT < 5 x institutional ULN in the presence of bone/liver metastases
* Serum creatinine (Cr) within ULN

  * Patients with Cr > ULN must have a Cr clearance of > 60 mL/min
* Testosterone 50 ng/mL or lower if a patient is receiving an LHRH agonist

  * No testosterone testing is required for men who have undergone surgical orchiectomy
* Fertile patients must agree to abstinence or some adequate form of contraception
* No patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs the ability to swallow AZD0530 tablets
* No history of uncontrolled or unstable cardiac dysrhythmia
* No resting ECG with measurable QTc interval of > 480 msec at 2 or more time points within a 24-hour period
* No evidence of interstitial lung disease (bilateral, diffuse, parenchymal lung disease)

  * A high-resolution CT of the chest will be required during screening
* No evidence of severe or uncontrolled systemic conditions (e.g., severe hepatic impairment) or current unstable or uncompensated respiratory or cardiac conditions which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol
* No patients with a known immunodeficiency syndrome
* No patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD0530
* No patients receiving any other investigational agents
* Previous AZD0530 exposure is allowed provided that the patient did not show radiographic progression during treatment
* Patients receiving non-steroidal anti-androgens (e.g., flutamide) or other hormonal treatment (such as ketoconazole, abiraterone, or TAK-700) must have stopped these drugs at least 28 days prior to enrollment for flutamide or ketoconazole, or at least 42 days prior to enrollment for bicalutamide or nilutamide, and the patients must have demonstrated progression of disease since the agents were suspended
* Patients should be at least 2 weeks away from previous chemotherapy, surgery, or radiotherapy
* No unresolved toxicity from previous treatments that are CTCAE grade 2 from previous anti-cancer therapy (except alopecia)
* Patients who are currently on zoledronic acid (Zometa) or other bisphosphonate therapy are eligible provided that they have been on therapy at least 6 weeks prior to participation

  * Increases in bisphosphonate dosing will not be allowed (i.e., starting within 6 weeks or changing from every 3-month to every 1-month dosing)
* Use of specifically prohibited CYP3A4-active agents or substances are not permitted during protocol treatment, and patients who must continue treatment with these agents are not eligible

  * Prohibited drugs should be discontinued 7 days prior to the administration of the first dose of AZD0530 and for 7 days following discontinuation of AZD0530 (unless otherwise specified)
* No concurrent use of non-FDA approved medications

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-12; Primary Completion 2012-09 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stadler, Principal Investigator — University of Chicago
Locations (15):
- United States (15):
  - University of Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - M D Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Women's Health Center, Madison, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Saracatinib): Patients receive 175 mg oral saracatinib once daily on days 1-28.
- Arm II (Placebo): Patients receive oral placebo once daily on days 1-28.
Period: Enrollment Phase
Arm/Group | Arm I (Saracatinib) | Arm II (Placebo)
Started | 33 | 0
Completed | 31 (Two patients signed consent but did not proceed to treatment.) | 0
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Lead-in Phase
Arm/Group | Arm I (Saracatinib) | Arm II (Placebo)
Started | 31 | 0
Completed | 8 (12 patients had radiographic progression, 8 clinical progression, 2 toxicity, 1 withdrawal.) | 0
Not Completed | 23 | 0
Not completed — Lack of Efficacy | 20 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Randomized Phase
Arm/Group | Arm I (Saracatinib) | Arm II (Placebo)
Started | 3 (3 of 8 patients randomized to saracatinib.) | 5 (5 of 8 patients randomized to placebo.)
Completed | 3 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients entering lead-in phase.
Groups:
- Arm I (Saracatinib): Patients receive 175 mg oral saracatinib once daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I (Saracatinib)
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 71 [48 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Duration of Stable Disease. (Time to Disease Progression by CT and/or Bone Scan or Clinical Progression.)
Description: Time to progression will be assessed using the Kaplan-Meier method and compared between groups via Wilcoxon rank-sum test.
Time Frame: Up to 6 months.
Population: Two patients in the placebo arm censored at 12 and 17 weeks, respectively.
Measure: Median (Full Range); unit: weeks
Arm/Group | Arm I (Saracatinib) | Arm II (Placebo)
Number analyzed (Participants) | 3 | 5
weeks | 18 [17 to 19] | 12 [9 to 17]
Statistical Analysis 1: Comparison: Arm I (Saracatinib) vs Arm II (Placebo); Test type: Superiority or Other; p = 0.20, Log Rank

2. Secondary Outcome: Toxicity and Incidence of Adverse Events
Description: Percentage of patients with grade 4 toxicity.
Time Frame: Up to 6 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Saracatinib) | Arm II (Placebo)
Number analyzed (Participants) | 3 | 5
percentage of participants | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 52.2]

3. Secondary Outcome: Toxicity and Incidence of Adverse Events.
Description: Percentage of patients who discontinued therapy due to toxicity.
Time Frame: Up to 6 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Saracatinib) | Arm II (Placebo)
Number analyzed (Participants) | 3 | 5
percentage of participants | 0.0 [0.0 to 70.8] | 20.0 [0.5 to 71.6]

4. Secondary Outcome: Correlation of Molecular Profile With Clinical Outcomes
Description: Study terminated after randomization of only 8 subjects. Correlative data not analyzed.
Time Frame: Up to 2 years
Arm/Group | Arm I (Saracatinib) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months (lead-in phase); up to 2 months (randomized phase).
Groups:
- Saracatinib, Lead-in Phase; Saracatinib, Randomized Phase: Patients receive 175 mg oral saracatinib once daily on days 1-28.
- Placebo, Randomized Phase: Patients receive placebo once daily on days 1-28.
Arm/Group | Saracatinib, Lead-in Phase | Saracatinib, Randomized Phase | Placebo, Randomized Phase
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/3 | 1/5
Other Adverse Events (participants affected / at risk) | 29/31 | 3/3 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saracatinib, Lead-in Phase (N=31) | Saracatinib, Randomized Phase (N=3) | Placebo, Randomized Phase (N=5)
Anemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saracatinib, Lead-in Phase (N=31) | Saracatinib, Randomized Phase (N=3) | Placebo, Randomized Phase (N=5)
Fatigue (General disorders) | 12 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 13 | 1 | 1
Nausea (Gastrointestinal disorders) | 9 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 7 | 0 | 0
Vomiting (Gastrointestinal disorders) | 9 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 8 | 0 | 0
Constipation (Gastrointestinal disorders) | 8 | 0 | 1
Creatinine increased (Renal and urinary disorders) | 4 | 0 | 0
Edema (General disorders) | 4 | 0 | 0
Fever (General disorders) | 5 | 0 | 0
Hematuria (Renal and urinary disorders) | 4 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0
Alkaline phosphatase increased (Investigations) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Confusion (Psychiatric disorders) | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 2 | 0 | 0
Neuropathy-sensory (Nervous system disorders) | 3 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 1 | 0
Pain (General disorders) | 7 | 1 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less